CLINICAL TRIAL: NCT01417013
Title: A Comparative Efficacy of SYSTANE® ULTRA vs Optive™ in Improving Tear Film Break-up Time
Brief Title: Comparative Efficacy of SYSTANE® ULTRA vs Optive™ in Improving Tear Film Break-up Time
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-10-07
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: Dry eye or lubricant eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Ultra (Active Comparator): Systane Ultra Lubricant Eye Drops
  Interventions: Other: Systane Ultra
- Optive (Active Comparator): Optive Lubricant eye drops
  Interventions: Other: Optive

INTERVENTIONS:
Other: Systane Ultra — Lubricant Eye Drops
  Other Names: Systane Ultra Lubricant Eye Drops
  Arms: Systane Ultra
Other: Optive — Lubricant eye drops
  Other Names: Optive Lubricant eye drops
  Arms: Optive

SUMMARY:
The primary objective of this study is assess the Tear Film break-up time (TBUT) in mild to moderate dry eye subjects.

DETAILED DESCRIPTION:
The primary objective of this study is assess the tear film break-up time in mild to moderate dry eye subjects.

ELIGIBILITY:
Inclusion Criteria:

* Corrected VA of 0.6 LogMar or better OU

Exclusion:

* Topical ocular medication use
* Presence of Ocular conditions (blepharitis, conjunctival infections, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
TBUT | 14 Days
  Tear Film break-up time